CLINICAL TRIAL: NCT01656473
Title: CIHR Team in Innovations in Child and Youth Concurrent Disorders: Service Delivery and Treatment Subproject
Brief Title: Evaluating the Effectiveness of Motivational Interviewing and a Dialectical Therapy Skills- Based Intervention for Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Children's Hospital of Eastern Ontario (Other); The Royal Ottawa Mental Health Centre (Other); Youth Services Bureau of Ottawa (Unknown)
Responsible Party: Principal Investigator, Shelley McMain, Head, Personality Disorders Treatment, Research and Capacity Building, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 069-2011
Record Dates: First submitted 2012-01-11; First posted 2012-08-03 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Concurrent Disorders
Keywords: Concurrent Disorders; Adolescents; Motivational Interviewing; Dialectical Behaviour Therapy; Caregiver Burden
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MI and DBT (Experimental): Individual Motivational Interview session followed by 12-week Dialectical Behaviour Therapy skills group
  Interventions: Other: MI and DBT

INTERVENTIONS:
Other: MI and DBT — One individual session of Motivational Interview followed by 12 weeks of Dialectical Behaviour Therapy group skills training
  Other Names: Integrated individual and group treatment
Other: MI and DBT — Individual Motivational Interview session plus 12-week Dialectical Behaviour Therapy skills group

SUMMARY:
The purpose of this study is to evaluate the preliminary effectiveness and feasibility of an integrated treatment approach for youth with concurrent disorders. The combined intervention will include individual sessions of Motivational Interviewing, followed by inclusion in a Dialectical Behaviour Therapy skills-based group.

The following main hypotheses will be examined:

1. Youth with CD who receive an MI intervention will show increased motivation and readiness to change from pre to post MI intervention.
2. Youth with CD who participate in a DBT intervention (orientation session followed by 12-week DBT skills training group)will show reductions in substance use and improvements in mental health, coping and affect regulation between pre to post treatment. The investigators expect that these treatment gains will be maintained at three-month follow-up.

DETAILED DESCRIPTION:
For this study, the investigators want to treat adolescents with concurrent disorders. Eligible subjects will be invited to participate in the combined intervention described in detail below.

In order to determine eligibility, designated research staff will conduct a phone screen interview with interested youth (ages 14 - 18). Candidates will be asked questions about their current mental health and substance use status. Based on the information obtained in this interview, those youth who report co-occurring mental health and substance use problems will be asked to complete three internet-based self-report questionnaires using a designated link and unique identification numbers. Once the information from this assessment is collected and scored by research personnel, those candidates who meet the criteria for this study will be asked to participate in the remaining portion of the study. These subjects will be required to meet with the research assistant in person to complete a computer-based self-administered structured diagnostic interview and self-report questionnaires.

If eligible and interested, subjects will be asked to meet with a therapist for one individual session of MI. These sessions will assess subjects' readiness to engage in treatment, and help identify treatment goals and any barriers that may make treatment difficult.

After these sessions, subjects will be invited to attend a DBT-focused orientation prior to joining the 12-week skills group. The investigators expect to have approximately 8 youth in each group and each session will run for 2 hours, weekly. The purpose of these group sessions is to learn skills that will help subjects cope in healthier ways. The following skills will be taught: (1) interpersonal effectiveness; (2) emotion regulation; (3) distress tolerance: and (4) mindfulness. The use of skills will be geared to addressing substance use problems and other mental health issues (e.g. anxiety, depression, self-harm, etc.).

Participants will be asked to complete questionnaires at the following time-points: screening, baseline, post-MI (2 weeks), mid-DBT (8 weeks), post-DBT (14 weeks), and at 14 weeks follow-up. Participants will be offered financial compensation upon completion of each assessment package.

ELIGIBILITY:
Inclusion criteria:

* age 14 to 18 years (inclusive);
* literacy in English;
* significant substance abuse problems indicated by a score in the problematic range on either the AUDIT (4 or above) or the DAST-A (6 or above);
* significant mental health problems as indicated by a score in the clinical range on at least one subscale of the YSR (T-score 65 or over);
* informed consent to participate in study;
* participation in regular case management or counselling (at least twice per month)1.

Exclusion criteria:

* history of schizophrenia or other psychotic disorder,
* evidence of an organic brain syndrome or severe intellectual disability;
* family members who are participating in the family intervention

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2012-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
(1) Substance Use: Teen Addiction Severity Index and; (2) Mental Health Symptoms: Youth Self-Report | Change from Baseline in Teen Addiction Severity Index and Youth Self-report at 2weeks, 8 weeks, 14 weeks, and 28 weeks
  Outcome measures to assess changes in mental health and substance use status.

SECONDARY OUTCOMES:
University of Rhode Island Change Assessment; Rutger's Alcohol Problem Index; Social Adjustment Scale-Adolescent Report; Difficulties in Emotion Regulation; Centre for Epidemiologic Studies in Depression | Change from Baseline in University of Rhode Island Change Assessment, Rutger's Alcohol Problem Index, Difficulties in Emotion Regulation, Social Adjustment Scale-Adolescent Report, Centre for Epidemiologic Studies in Depression at 2, 8, 14, and 28weeks
  In addition to outcome measurements for youth participants, adult caregivers will also be asked to complete two outcome measures: Stress Index of Parents of Adolescents; Child Behavior Checklist

CONTACTS AND LOCATIONS:
Overall Officials: Shelley McMain, PhD., Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital, fully affiliated with the University of Toronto, and a PAHO/WHO Collaborating Centre — http://www.camh.net/research